CLINICAL TRIAL: NCT04511312
Title: Management and Outcomes of Perioperative Care Among European Diabetic Patients: (MOPED): A Prospective Observational, International Cohort Study
Brief Title: Management and Outcomes of Perioperative Care Among European Diabetic Patients
Status: Recruiting | Type: Observational
Sponsor: European Society of Anaesthesiology (Other)
Responsible Party: Sponsor
Other Study IDs: MOPED
Record Dates: First submitted 2020-07-28; First posted 2020-08-13 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus; Postoperative Complications
Keywords: Diabetes Mellitus; Surgery; Postoperative complications
MeSH Terms: conditions — Diabetes Mellitus; Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The incidence of diabetes is increasing globally, including within Europe. There is an estimated 20million diabetic patients in Europe, which is likely to increase, thereby adding to societal demands on European health services. Diabetic patients are more likely to have surgical interventions than the general population. There are plausible pathophysiology and clinical mechanisms that diabetics are at increased risk of postoperative complications. When postoperative complications occur in the general population, they increase mortality or increase risk of major adverse cardiovascular events (Myocardial Infarction, Cerebrovascular Accident, Pulmonary embolism) at 30-days and up to one year later. In addition, diabetes is an independent risk factor for surgical site infections.

There is variation in practice guidelines in different countries in the perioperative management of diabetic patients undergoing major surgery, but this has not been documented on a large scale. Given the multiplicity of guidelines and differing recommendations, it is unsurprising that variability of 'real-world' clinical practice with regard to perioperative management of oral antihyperglycemic medications and insulin therapy has been noted in audits such as the National Confidential Enquiry into Patient Outcome and Death (NCEPOD).

Further, although it is recognised that diabetic patients are at increased risk of postoperative complications, this has not been recently evaluated, especially in light of ongoing developments in perioperative care, such as Enhanced Recovery Programmes. While a quality improvement intervention study has shown that maintaining tight preoperative glycaemic control improves postoperative glycaemic control, it is not known if this reduces postoperative morbidity overall. Further, whether certain anaesthetic techniques may be associated with better or worse outcomes after major non-cardiac surgery is unknown.

DETAILED DESCRIPTION:
see brief summary

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients (all classes except gestational diabetes) undergoing surgery (defined as requiring any general anaesthesia technique or any specific regional anaesthetic technique or a combination)
* Ambulatory, elective or emergency surgery and patients who receive postoperative care in intensive care or high dependency units will be included.

Exclusion Criteria:

* Patients who are not diabetic
* Patients with gestational diabetes
* Patients undergoing minor surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: General population
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Days at Home at 30 Days after surgery (DAH-30) | 30 days
  Number of days at home in the 30 days post surgery

SECONDARY OUTCOMES:
Comprehensive Complications Index (CCI) score, based on Clavien-Dindo scale; | Day 30
  Minimum score 0; Maximum score 100. Higher score indicates worse complications
Quality of Recovery QoR-15 measuring quality of recovery on Day 1 only | Day 1
  Minimum score 0; Maximum score 150. Higherscore indicates better recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- Mater University Hospital, Dublin, Ireland

REFERENCES:
- [Derived] Buggy DJ, Nolan R, Coburn M, Columb M, Hermanides J, Hollman MW, Zarbock A. Protocol for a prospective, international cohort study on the Management and Outcomes of Perioperative Care among European Diabetic Patients (MOPED). BMJ Open. 2021 Sep 6;11(9):e044394. doi: 10.1136/bmjopen-2020-044394. PMID 34489264